CLINICAL TRIAL: NCT01156246
Title: An Open Label, Randomized, Two-period, Crossover Study to Assess the Effect of Food on Fixed Dose Combination Dapagliflozin/Metformin Tablet (5 mg/1000 mg) in Healthy Male and Female Volunteers
Brief Title: Study to Assess the Effect of Food on Combination Dapagliflozin/Metformin Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1691C00005
Record Dates: First submitted 2010-06-28; First posted 2010-07-02 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Healthy volunteers; Dapagliflozin; Diabetes Type 2; Food interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dapagliflozin/metformin tablet, high fat, high calorie breakfast day 1, visit 2, 7-14 days wash-out, Dapagliflozin/metformin tablet, fasting conditions day 1, visit 3.
  Interventions: Drug: Dapagliflozin/Metformin
- 2 (Experimental): Dapagliflozin/metformin tablet, fasting conditions day 1, visit 2, 7-14 days wash-out, Dapagliflozin/metformin tablet, high fat, high calorie breakfast day 1, visit 3.
  Interventions: Drug: Dapagliflozin/Metformin

INTERVENTIONS:
Drug: Dapagliflozin/Metformin — oral fixed dose combination tablet 5 mg Dapagliflozin / 1000 mg Metformin given on day 1 at visit 2 and 3.

SUMMARY:
The purpose of this study is to determine whether treatment with a fixed dose combination dapagliflozin/metformin tablet is affected by food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI 18-30 kg/m2

Exclusion Criteria:

* History of clinically significant illness.
* History of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To assess the effect of food on the pharmacokinetics of dapagliflozin and metformin. | Serial PK sampling will be done on Days 1-4 at visit 2 and 3.
  primary - single dose Cmax, AUCinf, AUC(0-t) of dapagliflozin and metformin.. secondary - single dose tmax, t1/2 of dapagliflozin and metformin

SECONDARY OUTCOMES:
To examine the safety and tolerability of the fixed-dose combination tablet of dapagliflozin and metformin. | ECG at screening and follow-up. BP/pulse at screening, once daily during residential period and at follow-up. Clinical chemistry, haematology, and urine analyses at screening, day-1, day 4, and at follow-up.
  Vital signs (blood pressure and heart rate), electrocardiogram, laboratory safety data (clinical chemistry, haematology and urinalysis), adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB, Varvsgatan 53, SE-972 33 Luleå, Sweden; Wolfgang Kühn, Principal Investigator — Quintiles AB, Global Phase I Services, Strandbodgatan 1, SE-753 23 Uppsala, Sweden; Mirjana Kujacic, Study Chair — AZ Global Clinical Development, Pepparedsleden 1, 431 83 Mölndal, 431 83 Mölndal
Locations (1):
- Research Site, Luleå, Sweden